CLINICAL TRIAL: NCT03801369
Title: A Phase II, Open-Label, Study of Olaparib in Combination With Either Durvalumab (MEDI4736), Selumetinib or Capivasertib, or Ceralasertib Monotherapy in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: Olaparib in Combination With Either Durvalumab, Selumetinib, or Capivasertib or Ceralasertib Alone in Treating Patients With Metastatic Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of funding
Sponsor: Gordon Mills, MD, PhD (Other)
Collaborators: AstraZeneca (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor-Investigator, Gordon Mills, MD, PhD, IND Holder, OHSU Knight Cancer Institute
Organization: OHSU Knight Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018504; NCI-2019-00388 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018504 (Other: OHSU Knight Cancer Institute); STUDY00028065 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; capivasertib; ceralasertib; durvalumab; Immunoglobulin G; Disulfides; olaparib; AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (olaparib, durvalumab) (Experimental): Patients receive olaparib PO BID on days 1-28 of each cycle and durvalumab intravenously (IV) over 1 hour on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.
  Interventions: Procedure: Biopsy; Biological: Durvalumab; Drug: Olaparib; Other: Quality-of-Life Assessment
- Arm II (olaparib, selumetinib) (Experimental): Patients receive olaparib PO BID on days 1-28 of each cycle and selumetinib PO BID on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.
  Interventions: Procedure: Biopsy; Drug: Olaparib; Other: Quality-of-Life Assessment; Drug: Selumetinib
- Arm III (olaparib, capivasertib) (Experimental): Patients receive olaparib PO BID on days 1-28 of each cycle and capivasertib PO BID 4 days on and 3 days off of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.
  Interventions: Procedure: Biopsy; Drug: Capivasertib; Drug: Olaparib; Other: Quality-of-Life Assessment
- Arm IV (ceralasertib) (Experimental): Patients receive ceralasertib PO BID on days 1-14 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.
  Interventions: Procedure: Biopsy; Drug: Ceralasertib; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Capivasertib — Given PO (orally)
  Other Names: AZD5363
  Arms: Arm III (olaparib, capivasertib)
Drug: Ceralasertib — Given PO (orally)
  Other Names: AZD6738
  Arms: Arm IV (ceralasertib)
Biological: Durvalumab — Given IV (infusion)
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
  Arms: Arm I (olaparib, durvalumab)
Drug: Olaparib — Given PO (orally)
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
  Arms: Arm I (olaparib, durvalumab); Arm II (olaparib, selumetinib); Arm III (olaparib, capivasertib)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Selumetinib — Given PO (orally)
  Other Names: ARRY-142886; AZD6244; MEK Inhibitor AZD6244
  Arms: Arm II (olaparib, selumetinib)

SUMMARY:
This phase II study assesses the efficacy of the combination of olaparib with durvalumab, selumetinib, or capivasertib or ceralasertib alone in the treatment of patients with metastatic triple negative breast cancer (TNBC). Olaparib may stop growth of tumor cells by inhibiting some of the enzymes (ADP ribose polymerase [PARP]) needed for cell growth. Durvalumab, a monoclonal antibody, inhibits the growth and spread of tumors by stimulating the patient's antitumor immune response. Selumetinib, capivasertib, and ceralasertib are inhibitor drugs that may stop the growth of tumor cells by blocking some of the enzymes (MEK, AKT, ATR) needed for cell growth. Giving olaparib together with durvalumab, selumetinib, or capivasertib or giving ceralasertib alone may provide an effective method to treat patients with metastatic triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess overall response to treatment.

SECONDARY OBJECTIVES:

I. Assess participant benefit from treatment. II. Determine the time to disease progression following response to study therapy.

III. Determine time to first disease progression or death of participants enrolled on the study.

IV. Determine survival of participants enrolled on the study. V. Assess safety and tolerability of the proposed therapy.

EXPLORATORY OBJECTIVES:

I. To assess a change in quality of life (QOL) as measured by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) in each treatment arm.

II. To assess a change in QOL as measured by Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23) in each treatment arm.

III. Examine response rates depending on tumor characteristics. IV. Identify predictive biomarkers of sensitivity to therapy. V. Identify emerging mechanism of resistance to therapy. VI. Determine changes in tumor cells and the tumor microenvironment induced by PARP inhibitors.

OUTLINE: This is an open-label, multi-arm phase II study of olaparib in combination with durvalumab, selumetinib, or capivasertib, or ceralasertib monotherapy.

LEAD IN: Patients with biopsy proven TNBC undergo a pre-treatment biopsy. At the 2 week mark, patients then undergo a repeat on-treatment biopsy. Patients also receive olaparib orally (PO) twice daily (BID) on days 1-28 for one cycle. Treatment repeats every 28 days for up to 1 cycle in the absence of disease progression or unacceptable toxicity.

Patients are then assigned to 1 of 4 arms based on predefined molecular tumor characteristics.

ARM I: Patients receive olaparib PO BID on days 1-28 of each cycle and durvalumab intravenously (IV) over 1 hour on day 1 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.

ARM II: Patients receive olaparib PO BID on days 1-28 of each cycle and selumetinib PO BID on days 1-28 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.

ARM III: Patients receive olaparib PO BID on days 1-28 of each cycle and capivasertib PO BID 4 days on and 3 days off of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.

ARM IV: Patients receive ceralasertib PO BID on days 1-14 of each cycle. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit from treatment may, at the investigator's discretion and in the absence of disease progression or unacceptable toxicity, continue on therapy beyond the planned 13 cycles.

At the completion of all on-study procedures, patients are followed up every 6 months for disease and survival outcomes up to 1 year. Patients will be asked to submit an optional tumor biopsy in the event of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participants are >= 18 years old at time of informed consent.
* Metastatic TNBC, as defined by:

  * Estrogen receptor (ER) and progesterone receptor (PR) negative as defined as ER < 10% and PR < 10% by immunohistochemistry according to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines for hormone receptor testing
  * HER2 non-amplified per ASCO/CAP guidelines, defined as:

    * IHC score 0/1+
    * IHC 2+ and in situ hybridization (ISH) non-amplified with a ratio of HER2 to CEP17 < 2.0, and if reported, average HER2 gene copy number < 4 signals/cells; or
    * ISH non-amplified with a ratio of HER2 to CEP17 <2.0, and if reported, average HER2 gene copy number < 4 signals/cells
* Participants with or without germline BRCA mutated TNBC are eligible for study participation
* Participants must have at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 that is amenable to biopsy
* Prior therapies for metastatic breast cancer

  * Frontline patients who have not received prior systemic therapy for metastatic breast cancer are eligible
  * Patients who have received =< 2 prior chemotherapy regimens for metastatic breast cancer are eligible
* Participants must have fully recovered from the acute toxic effects of all prior treatment to grade 1 or less, except alopecia which is allowed
* Participants must have a life expectancy >= 16 weeks
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Participant must consent to undergo a pre-treatment screening biopsy for enrollment and subsequent biomarker analyses
* Participants must consent to undergo one mandatory on-study tumor biopsy following a 2-week induction treatment of olaparib. A second on-study biopsy at time of disease progression is optional, but not mandatory
* Participants must not have received previous treatment with PARP inhibitors, including olaparib
* Hemoglobin >= 10.0 g/dL (measured within 28 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (measured within 28 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 28 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5 x ULN (measured within 28 days prior to administration of study treatment)
* Participants must have creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test (measured within 28 days prior to administration of study treatment)
* Participants of childbearing potential must have a negative urine or serum pregnancy test within 28 days of study treatment and confirmed on Day 1 prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants of childbearing potential agree to use adequate methods of contraception, upon signing of informed consent through:

  * 6 months after the last dose with olaparib,
  * 3 months after the last dose with durvalumab,
  * 1 week after the last dose with selumetinib,
  * 1 month after the last dose with capivasertib,
  * 1 month after the last dose with ceralasertib.
* Participants of childbearing potential are those who are not proven postmenopausal. Postmenopausal is defined as:

  * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
  * Radiation-induced oophorectomy with last menses >1 year ago
  * Chemotherapy-induced menopause with >1 year interval since last menses
  * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Sperm-producing participants must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant partner or with an individual of childbearing potential. Partners of sperm-producing participants should also use a highly effective form of contraception if they are of childbearing potential

  * Sperm-producing participants assigned to receive capivasertib must use a condom during treatment and for 4 months after the last dose of capivasertib when having sexual intercourse with a pregnant partner or with an individual of childbearing potential

Exclusion Criteria:

* Any concurrent anticancer treatment

  * Individuals in the follow-up phase of a prior investigational study may participate as long as it has been 4 weeks since last dose of the previous investigational agent or device
  * Concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replacement therapy) is allowed
* Participant's with tumors showing androgen receptor (AR) >= 80% by immunohistochemistry are excluded
* Other malignancy unless curatively treated with no evidence of disease for >= 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma. Participants with a personal history of treated early stage breast cancer whose natural history or treatment does not have the potential to interfere with the safety or efficacy endpoints of the trial, per investigator assessment, are eligible
* Participants with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Participant received prior anticancer therapy such as targeted therapies, or systemic chemotherapy or radiation (except for palliative reasons) within the past 3 weeks, or 5 half-lives, whichever is shorter, prior to first day of treatment
* Participants with known active central nervous system (CNS) metastases and/or carcinomatous meningitis

  * Patients with brain metastases may participate provided they do not have symptomatic uncontrolled disease. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. (note: a scan to confirm the absence of brain metastases is not required)
  * Patients with spinal cord compression are not eligible unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
  * Patients with carcinomatous meningitis are not eligible
* Concomitant use of known strong CYP3A inhibitors (e.g., ketoconazole, posaconazole), or strong CYP3A inducers (e.g., phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study intervention treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Patients that are immunocompromised, including those with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness are not eligible for participation

  * Note: HIV-infected participants on effective anti-retroviral therapy with undetectable viral load for >= 6 months are eligible for this trial provided that there is minimal interactions or overlapping toxicity of the antiretroviral therapy with their study intervention. Refer to drug-specific exclusion criteria for additional considerations
* Patients with known active hepatitis (i.e. hepatitis B or C). Refer to drug-specific exclusion criteria for additional considerations

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result
  * Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA. Those with a positive HCV PCR will be excluded
* Participants unable to swallow orally administered medication and participants with gastrointestinal disorders likely to interfere with absorption of the study medication
* Participants with visceral crisis defined as severe organ dysfunction as assessed by signs and symptoms, laboratory studies, and rapid progression of disease
* Active infection requiring systemic antibiotic therapy. Participants requiring systemic antibiotics for infection must have completed therapy before treatment is initiated
* Participants considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric illness/social situation that prohibits obtaining informed consent
* Resting electrocardiography (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, corrected QT interval by Fridericia's correction formula (QTcF) prolongation > 500 ms, electrolyte disturbances, etc.), or participants with congenital long QT syndrome
* Participants with a history of hypersensitivity reactions to study agent, olaparib, or its excipients
* Participant is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Sperm-producing participants are prohibited from donating sperm upon signing of informed consent through:

  * 3 months following last dose with olaparib
  * 4 months following last dose with capivasertib
  * 6 months following last dose with ceralasertib
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* DRUG-SPECIFIC EXCLUSION CRITERIA: The following criteria require consideration for participant eligibility to one or more of the available treatment arms. Participant eligibility may be assessed at the time of initial screening or as part of the on-study assignment to a specific treatment arm
* DURVALUMAB EXCLUSION CRITERIA: Participant has received prior immunotherapy with anti-PD-L1, including durvalumab anti-PD-1, anti-CTLA4 or similar drugs in the metastatic setting
* DURVALUMAB EXCLUSION CRITERIA: Participants may have received prior immunotherapy in the adjuvant setting, provided

  * No documented disease progression on immunotherapy
  * Treatment with immunotherapy was >1 year from enrollment on study
* DURVALUMAB EXCLUSION CRITERIA: Participant has evidence of interstitial lung disease or active non-infectious pneumonitis
* DURVALUMAB EXCLUSION CRITERIA: Major surgery within 2 weeks of starting study treatment and participants must have recovered from any effects of any major surgery

  * Note: Local surgery of isolated lesions for palliative intent is acceptable per investigator discretion
* DURVALUMAB EXCLUSION CRITERIA: Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus

  * Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
  * Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
  * Those with controlled human immunodeficiency virus (HIV) are eligible, provided that:

    * Baseline CD4+ T-cell count is >= 200 cells/mm^3, and
    * HIV plasma viral load is < 60 copies/ml
* DURVALUMAB EXCLUSION CRITERIA: History of active primary immunodeficiency
* DURVALUMAB EXCLUSION CRITERIA: Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication)
* DURVALUMAB EXCLUSION CRITERIA: Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Participants with vitiligo or alopecia
  * Participants with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Participants without active disease in the last 5 years may be included but only after consultation with the study physician
  * Participants with celiac disease controlled by diet alone
* DURVALUMAB EXCLUSION CRITERIA: History of allogenic bone marrow transplant or double umbilical cord blood transplantation
* DURVALUMAB EXCLUSION CRITERIA: Participants must not have received live vaccines within 30 days prior to the first dose of

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Mills, MD, PhD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Sun C, Fang Y, Labrie M, Li X, Mills GB. Systems approach to rational combination therapy: PARP inhibitors. Biochem Soc Trans. 2020 Jun 30;48(3):1101-1108. doi: 10.1042/BST20191092. PMID 32379297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Started | 24 | 0 | 0 | 0
Completed | 24 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Arms II - IV.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Olaparib, Durvalumab) | Arm II (Olaparib, Selumetinib) | Arm III (Olaparib, Capivasertib) | Arm IV (Ceralasertib) | Total
Number analyzed (Participants) | 24 | 0 | 0 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  |  | 0
  Between 18 and 65 years | 20 |  |  |  | 20
  >=65 years | 4 |  |  |  | 4
Age, Continuous [Mean (Full Range); unit: Years] | 54 [25.3 to 78.9] |  |  |  | 54 [25.3 to 78.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 |  |  |  | 24
  Male | 0 |  |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 24 |  |  |  | 24
  Unknown or Not Reported | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  | 0
  Asian | 0 |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  | 0
  Black or African American | 1 |  |  |  | 1
  White | 21 |  |  |  | 21
  More than one race | 0 |  |  |  | 0
  Unknown or Not Reported | 2 |  |  |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 |  |  |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Using the efficacy analysis set, the estimate of ORR will be measured independently for each treatment arm and reported with 95% exact confidence interval. Participants who, within their respective treatment arm, achieve a complete response (CR) or a partial response (PR) that is confirmed on a second scan at least 4 weeks later on the current protocol will be qualified as achieving a response, and will count towards the ORR measurement.
Time Frame: End of treatment (Up to 24 months)
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 21 | 0 | 0 | 0
Participants | 6 |  |  |

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: An estimate of CBR will be measured independently for each treatment arm and reported with 95% exact confidence interval. Participants who, within their respective treatment arm, achieve a CR, PR, or stable disease (SD) for at least 6 months on the current protocol will be qualified as deriving benefit from therapy, and will count towards the CBR measurement.
Time Frame: End of treatment (Up to 24 months)
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 21 | 0 | 0 | 0
Participants | 10 |  |  |

3. Secondary Outcome: Duration of Response (DOR)
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented taking as reference for progressive disease the smallest measurements recorded since the treatment started. The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented. If a participant dies, irrespective of cause, without documentation of recurrent or progressive disease beforehand, then the date of death will be used to denote the response end date.
Time Frame: End of treatment (Up to 24 months)
Reporting Status: Not Posted

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time after having completed at least one cycle of olaparib monotherapy to the first of either recurrence or relapse (anywhere in the body) or death at the time of last follow-up at 12-months. The estimated distribution of the PFS for each treatment will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available.
Time Frame: Progression or death (any cause) up to 1 year post treatment
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Mean (Full Range); unit: months
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 20 | 0 | 0 | 0
months | 4.8 [2.17 to 8.97] |  |  |

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time after having completed at least one cycle of olaparib monotherapy up to 6 months following the completion of on-study treatment to the date of death or last follow-up at 12 months. The estimated distribution of the OS for each treatment will be plotted using Kaplan Meier curves and reported with median survival and 95% confidence intervals if available.
Time Frame: Death (any cause) up to 1 year post treatment
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 24 | 0 | 0 | 0
months | 15.5 [7.85 to 18.1] |  |  |

6. Secondary Outcome: Incidence of Grade 3+ Acute Toxicity
Description: Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The incidence of having grade 3+ acute toxicity will be determined for participants with triple negative breast cancer (TNBC) that received at least one dose of olaparib and/or durvalumab., selumetinib, capivasertib, or ceralasertib. The 95% confidence interval will be reported with the point estimate of toxicity rate.
Time Frame: Up to 3 months post treatment
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Number; unit: occurrences
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 24 | 0 | 0 | 0
occurrences | 46 |  |  |

7. Other Pre Specified Outcome: Change in Quality of Life (QOL) as Measured by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: The QOL measures will be summarized and presented over time graphically using box and spaghetti plots, in addition to summary tables. Mixed effect model will be further used to analyze the longitudinal data. For each instrument, the analysis will include all cycles for which at least 25% of participants in each arm that have an assessment. QLQC30 is a 30-item measure and yields scores for 5 functional scales (physical, role, cognitive, social, and emotional), 3-symptom scales (nausea, pain, and fatigue), a global health and QOL scale, and perceived financial impact of treatment. QLQC30 can distinguish patients according to performance status and is the most commonly used QOL instrument in oncology research. Data from the EORTC QLQ-C30 instrument will be scored as previously described by Aaronson et al.
Time Frame: Baseline to end of treatment (Up to 24 months)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in QOL as Measured by EORTC QLQBR23
Description: The QOL measures will be summarized and presented over time graphically using box and spaghetti plots, in addition to summary tables. Mixed effect model will be further used to analyze the longitudinal data. For each instrument, the analysis will include all cycles for which at least 25% of participants in each arm that have an assessment. QLQBR23 is a 23-item instrument that measures symptoms and side effects related to treatment, body image, sexuality, and future perspective specific to breast cancer patients. QLQBR23 has high internal consistency (Cronbach's a = 0.71-0.90), can distinguish between patients based on disease stage, performance status, treatment modality, or prior surgery, and is sensitive to change over time. The EORTC QLQ-BR23 data will be scored as described by the EORTC scoring manual.
Time Frame: Baseline to end of treatment (Up to 24 months)
Reporting Status: Not Posted

9. Secondary Outcome: Incidence of Grade 3+ Acute Toxicity
Description: as for outcome 6
Time Frame: Up to 3 months post treatment
Population: No participants were enrolled in Arm II - Arm IV.
Measure: Number; unit: participants
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
Number analyzed (Participants) | 24 | 0 | 0 | 0
participants | 16 |  |  |

ADVERSE EVENTS:
Time Frame: 6 years
Description: No participants were enrolled in Arm II - Arm IV.
Arm/Group | Arm I (olaparib, durvalumab) | Arm II (olaparib, selumetinib) | Arm III (olaparib, capivasertib) | Arm IV (ceralasertib)
All-Cause Mortality (participants affected / at risk) | 19/24 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/24 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 24/24 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (olaparib, durvalumab) (N=24) | Arm II (olaparib, selumetinib) (N=0) | Arm III (olaparib, capivasertib) (N=0) | Arm IV (ceralasertib) (N=0)
Motor Vehicle Accident (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (olaparib, durvalumab) (N=24) | Arm II (olaparib, selumetinib) (N=0) | Arm III (olaparib, capivasertib) (N=0) | Arm IV (ceralasertib) (N=0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 12 (40) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders (Eye disorders) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 22 (95) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions (General disorders) | 13 (29) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 10 (24) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 5 (16) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 9 (20) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 9 (15) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 15 (39) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 16 (40) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 7 (11) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 16 (49) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Surgical and Medical Procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03801369/Prot_SAP_001.pdf